CLINICAL TRIAL: NCT06945042
Title: The Impact of Systematic Financial Navigation in Acute Myeloid Leukemia "SF-NAV"
Brief Title: ONC-LEUK-2406: The Impact of Systematic Financial Navigation in Acute Myeloid Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); Swim Across America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00126844; ONC-LEUK-2406 (Other: Atrium Health)
Record Dates: First submitted 2025-03-27; First posted 2025-04-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Financial Navigation; Financial Toxicity
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic Financial Navigation (Other): Participants randomized to Arm A will initiate navigation as soon as feasibly possible after randomization but no later than 4 weeks from enrollment.
  The intervention will consist of systematic financial navigation with consistent screening and intervention on any financial related issues. The clinical trials staff will refer the participant to the appropriate services for personalized recommendations and assistance provided by Atrium Health personnel including financial navigators, nurse navigators. All the resources provided to the patient, including counseling, will be free of charge. Assessment will be performed once per month for 6 months.
  Interventions: Other: Arm A
- Standard of Care Financial Distress Intervention (Other): Participants randomized to Arm B will receive standard of care financial distress treatment including nurse navigation and pharmacy resources as soon as feasibly possible after randomization but no later than 4 weeks from enrollment.
  All patients randomized to the Standard of Care arm will have access to the financial distress resources (Financial Navigation and Nurse Navigation) as per current clinical policy which is per patient or clinician request. All the resources provided to the patient, including counseling, will be free of charge as per institutional policy.
  Interventions: Other: Arm B

INTERVENTIONS:
Other: Arm A — The intervention will consist of systematic financial navigation with consistent screening and intervention on any financial related issues. All patients randomized to the financial navigational group will be contacted by clinical trial staff assigned to the study to screen for financial needs. Based on the results of this assessment, the clinical trials staff will refer to the appropriate services for personalized recommendations and assistance provided by Atrium Health personnel including financial navigators, nurse navigators. All the resources provided to the patient, including counseling, will be free of charge. Assessment will be performed once per month for 6 months.
  Arms: Systematic Financial Navigation
Other: Arm B — All patients randomized to the Standard of Care arm will have access to the financial distress resources (Financial Navigation and Nurse Navigation) as per current clinical policy which is per patient or clinician request. Utilization of these resources will be tracked to assess and describe the per-protocol population. All the resources provided to the patient, including counseling, will be free of charge as per institutional policy.
  Arms: Standard of Care Financial Distress Intervention

SUMMARY:
The purpose of this research is to see how personal financial burden (financial toxicity) related to cancer affects the overall health and quality of life by evaluating the impact of systematic financial navigation in addition to standard financial distress interventions during cancer treatment.

DETAILED DESCRIPTION:
Financial navigation (FN) has been increasingly recognized as an important interventional tool with the potential to significantly mitigate the onset, severity, and duration of financial toxicity (FT). There have been several recent pilot studies in this area demonstrating the feasibility and effectiveness of this approach. With the suddenness of onset and high healthcare utilization of an acute leukemia diagnosis, financial navigation early in the disease course may represent an opportunity to reduce the financial distress burden of this disease and improve outcomes.

The investigators have chosen to conduct this as a randomized, controlled trial (RCT) evaluating the effect of financial navigation (FN) on the patient reported objective measurement of financial toxicity (FT) using the Comprehensive Score for Financial Toxicity (COST) measure. This 12-question measure has become the standard for financial toxicity (FT) quantification in the research setting and will allow for direct comparison between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an IRB-approved informed consent.
2. Age 18-64 years at the time of consent
3. Initial diagnosis of Acute Myeloid Leukemia (AML) per investigator Note: Date of initial diagnosis is the date of the bone marrow biopsy
4. Planned intensive induction chemotherapy Note: It is acceptable if chemotherapy has been initiated at the time of enrollment as long as it is within 30 days of therapy initiation
5. Ability to read and understand the English and/or Spanish language(s)
6. As determined by the enrolling investigator, ability of the participant to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Diagnosis of Acute Promyelocytic Leukemia
2. Unwilling to receive induction chemotherapy for AML
3. Previous treatment for hematologic malignancy
4. Prior allogeneic hematopoietic stem cell transplant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Self-reported financial toxicity as assessed by the total score of the COmprehensive Score Financial Toxicity (COST) assessment tool at 6 months after enrollment. | From the date of randomization up until six months
  For each participant, the total score of the COST at the 6-month assessment will be calculated. The total score is informed by 11 questions, each assessed on a 5-point scale of numerical values ranging 0 to 4, and the total score may range from 0 to 44 (where the lower score, the worse the financial well-being of the participant).
  Data of COST assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.

SECONDARY OUTCOMES:
Self-reported financial toxicity as assessed by the total score of the COmprehensive Score Financial Toxicity (COST) assessment tool at 3 months after enrollment. | From the date of randomization up until three months
  For each participant, the total score of the COST at the 3-month assessment will be calculated. The total score is informed by 11 questions, each assessed on a 5-point scale of numerical values ranging 0 to 4, and the total score may range from 0 to 44 (where the lower score, the worse the financial well-being of the participant).
  Data of COST assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported financial toxicity as assessed by the total score of the COmprehensive Score Financial Toxicity (COST) assessment tool at 12 months after enrollment. | From the date of randomization up until twelve months
  For each participant, the total score of the COST at the 12-month assessment will be calculated. The total score is informed by 11 questions, each assessed on a 5-point scale of numerical values ranging 0 to 4, and the total score may range from 0 to 44 (where the lower score, the worse the financial well-being of the participant).
  Data of COST assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported physical health as assessed by the total score of the Global Physical Health (GPH) as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) at 3 months after enrollment | From the date of randomization up until three months
  For each participant, the total score of the GPH measure at the 3-month assessment will be calculated. The total raw score is informed by four items and the total raw score may range from 4 to 20 (where the higher score represents more physical health). The total raw score will be standardized to the general population using the scale's published T-scores. The transformed T scores will be used in analyses and range from 16.2 to 67.7.
  Data of GPH assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported physical health as assessed by the total score of the Global Physical Health (GPH) as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) at 6 months after enrollment | From the date of randomization up until six months
  For each participant, the total score of the GPH measure at the 6-month assessment will be calculated. The total raw score is informed by four items and the total raw score may range from 4 to 20 (where the higher score represents more physical health). The total raw score will be standardized to the general population using the scale's published T-scores. The transformed T scores will be used in analyses and range from 16.2 to 67.7.
  Data of GPH assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported physical health as assessed by the total score of the Global Physical Health (GPH) as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) at 12 months after enrollment | From the date of randomization up until twelve months
  For each participant, the total score of the GPH measure at the 12-month assessment will be calculated. The total raw score is informed by four items and the total raw score may range from 4 to 20 (where the higher score represents more physical health). The total raw score will be standardized to the general population using the scale's published T-scores. The transformed T scores will be used in analyses and range from 16.2 to 67.7.
  Data of GPH assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported physical health as assessed by the total score of the Global Mental Health (GMH) as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) at 3 months after enrollment | From the date of randomization up until three months
  For each participant, the total score of the GMH measure at the 3-month assessment will be calculated. The total raw score is informed by four items and the total raw score may range from 4 to 20 (where the higher score represents more physical health). The total raw score will be standardized to the general population using the scale's published T-scores. The transformed T scores will be used in analyses and range from 21.2 to 67.6.
  Data of GPH assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported physical health as assessed by the total score of the Global Mental Health (GMH) as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) at 6 months after enrollment | From the date of randomization up until six months
  For each participant, the total score of the GMH measure at the 6-month assessment will be calculated. The total raw score is informed by four items and the total raw score may range from 4 to 20 (where the higher score represents more physical health). The total raw score will be standardized to the general population using the scale's published T-scores. The transformed T scores will be used in analyses and range from 21.2 to 67.6.
  Data of GPH assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported physical health as assessed by the total score of the Global Mental Health (GMH) as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) at 12 months after enrollment | From the date of randomization up until twelve months
  For each participant, the total score of the GMH measure at the 12-month assessment will be calculated. The total raw score is informed by four items and the total raw score may range from 4 to 20 (where the higher score represents more physical health). The total raw score will be standardized to the general population using the scale's published T-scores. The transformed T scores will be used in analyses and range from 21.2 to 67.6.
  Data of GPH assessments from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported gaps in care as assessed by the number of gaps of care reported in the Financial Navigation Intervention Compliance/Coping Survey at 3 months after enrollment | From the date of randomization up until three months
  For each participant, the total number of gaps of care reported in the Financial Navigation Intervention Compliance/Coping Survey at the 3-month assessment will be calculated. The total score is informed by 9 questions, each assessed as a binary response "Yes/No", where each response of "Yes" will be mapped to a numerical value of 1 and each "No" will be mapped to a numerical value of 0. The total sum will be calculated as the total score and the total score may range from 0 to 9 (where the higher score represents the most severe gaps in care assessed by the survey).
  Data from the Financial Navigation Intervention Compliance/Coping Survey from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported gaps in care as assessed by the number of gaps of care reported in the Financial Navigation Intervention Compliance/Coping Survey at 6 months after enrollment | From the date of randomization up until six months
  For each participant, the total number of gaps of care reported in the Financial Navigation Intervention Compliance/Coping Survey at the 6-month assessment will be calculated. The total score is informed by 9 questions, each assessed as a binary response "Yes/No", where each response of "Yes" will be mapped to a numerical value of 1 and each "No" will be mapped to a numerical value of 0. The total sum will be calculated as the total score and the total score may range from 0 to 9 (where the higher score represents the most severe gaps in care assessed by the survey).
  Data from the Financial Navigation Intervention Compliance/Coping Survey from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Self-reported gaps in care as assessed by the number of gaps of care reported in the Financial Navigation Intervention Compliance/Coping Survey at 12 months after enrollment | From the date of randomization up until twelve months
  For each participant, the total number of gaps of care reported in the Financial Navigation Intervention Compliance/Coping Survey at the 12-month assessment will be calculated. The total score is informed by 9 questions, each assessed as a binary response "Yes/No", where each response of "Yes" will be mapped to a numerical value of 1 and each "No" will be mapped to a numerical value of 0. The total sum will be calculated as the total score and the total score may range from 0 to 9 (where the higher score represents the most severe gaps in care assessed by the survey).
  Data from the Financial Navigation Intervention Compliance/Coping Survey from all randomized participants will inform this intent-to-treat analysis comparing scores between the arms.
Overall survival | From the date of randomization up until date of death or last known follow-up, assessed over 3 years.
  Overall survival is defined as the time interval from the date of diagnosis to the date of death from any cause, or the date of last known follow-up while on study.
  All randomized participants will inform this analysis.
Comparison of relapse-free survival All randomized participants will inform this analysis. | From the date of randomization up until date of relapse, death or last known follow-up, assessed over 3 years.
  Relapse-free survival is defined as the time interval from the completion of initial treatment (which may include induction and consolidation therapy) to the date of the first documented relapse of AML or death from any cause, whichever occurs first. A relapse is characterized by the re-emergence of leukemia cells in the bone marrow or peripheral blood; in absence of disease relapse, participants will be censored at the last follow-up visit where they were confirmed to be in complete remission without evidence of relapse. Relapse-free survival will be calculated for participants achieving complete response after initial treatment only.
Annualized count of acute care visits | From the date of randomization up until twelve months
  The annualized count of acute care visits, where acute care visits include all unplanned hospital admissions and unplanned emergency department visits was calculated for each participant as the total number of acute care visits normalized to an annual basis. Data of randomized will inform this intent-to-treat analysis comparing counts between the arms.
  All randomized participants will inform this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Knight, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Insitute, Charlotte, North Carolina, United States